CLINICAL TRIAL: NCT05356442
Title: Association of Tenodesis Grip Strength With Functional Hand Recovery in Patients With Cervical Spinal Cord Injury
Brief Title: Tenodesis Grip Strength With Functional Hand Recovery in Cervical Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/Lhr/22/0209 Amna Ali
Record Dates: First submitted 2022-04-28; First posted 2022-05-02 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury, pain ,tenodesis grip, strength
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal cord injury (SCI) is devastating event, the individual become significant burden on their family and society SCI is impairments of sensory, motor and autonomic functions. There is no proper cure and care after SCI, no proper assessment and treatment is present in under developed countries Cross sectional study design will be used and 75 patients included in this study. The population included age 21-55 years, both gender included, teraplegic with lesion level C5-C7, Mini Mental State of Examination ≥24, patient should be medically stable. The patient excluded with history of peripheral nerve lesion as brachial pluxes impairment. For assessment of hand function tools should be used tenodesis grip strength is assessed Graded Redefined Assessment of Strength sensibility and prehension (GRASSP test), and functional hand recovery assessed by jebsen_Taylor Hand function test (JTHFT_IT), hand dynamo meter for grip strength, Action Arm reach test for hand function and spinal cord independence measure will be used. Pearson correlation will be uses to find the association between hand grip strength and functional activities of hand. The collected data will be analyzed by using SPSS 23.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is important area for research, because of planning the services for the disabled and also decisions making for the prevention and control of SCI. Spinal cord injury (SCI) is a highly destructive and damaging condition with enormous financial, social, and personal costs. As, there is no known cure for SCI. so, primary prevention is a necessary. Due to high incidence of road traffic accidents, epidemiologic data concerning that, it is the specific causes of spinal cord injury and the other causes of spinal cord injury Traumatic including transport, fall, diving in shallow water, other may be non- traumatic including iatrogenic. So, the understanding of this is important due to preventive strategies and for planning better treatment and cure. The most devastating aspects of spinal cord injury are Quadriplegia because it is the impairment of arm and hand function, which badly affect the individual's level of independence. Improving arm and hand function has been reported to be a high priority for individuals with SCI.As, the hand function change with neurological level of lesion specially in cervical spinal cord injury. In which hand function is almost completely loss above C5 and below C7 cord lesion the upper limb functions almost preserved. The high priority is preserved hand function due to personal independence and improve the quality of life. Tenodesis function is used to facilitate the functional hand grasp and release by adjusting the position of wrist in tetraplagic peoples. When the wrist flexed, fingers and thumb open and when the wrist extended, fingers and thumb flexed into palm. It is possible for those who have wrist extension in grade 3 and no active movement of fingers Tenodesis grasp is useful for C6-C7 spinal cord injury because they have control on wrist movement and limited finger control. So they can easily grasp and release objects than those who have no or limited control over their hands. That is helpful for their ADLs. Functional hand recovery or hand strength in Quadriplegia is improved with repetitive active or passive ROM. The above and below the spinal level of lesion. Hand grip devices also used for improving the grip strength and hand function in SCI.According to searched data no study conducted to describe the association between the functional hand recovery with reference to neurological lesion level of cervical spinal cord injury and tenodesis grip strength. To find out the association between the tenodesis grip and functional hand recovery in patient with cervical spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age group is from 21 to 55 years.
* Both male and female
* Tetraplegic with neurological lesion level C5-C7
* Mini Mental State Examination ≥24
* Grade C and D will include in this study according to ASIA impairment scale
* Upper limb muscles in grade 0, 1, +1 according to modified Ashworth scale

Exclusion Criteria:

* Contracture of upper extremity with C5-C7 cervical SCI.
* Combined peripheral or central nervous system disease
* History of peripheral nerve lesion as brachial plexus impairment
* Previously known poly Neuropathy or sever cranio cerebral injury
* History of Fracture or any surgical procedure in hand area.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: SCI
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Graded Redefined Assessment of Strength Sensibility and Prehension (GRASSP) | 8 months
  GRASSP is a clinical research tool for sensory and motor impairment data of upper limb in cervical spinal cord injury. GRASSP have three components, first is sensibility domain test site is selected by dermatome, second is strength and tone domain in which muscle tested by myotomes and third is prehension domain in which segmental influence movement pattern
Jebsen-Taylor hand function test (JTHFT-IT) | 8 months
  JTHFT-IT is used in people with tetraplegia. This scale is used for assessment of arm and hand , including basic functions as moving objects in which turning and pick up small objects , lifting small objects and light weighted objects also grasp and release including complex functions as dress up and toileting. The maximum time for execution of seven items will be 14min since the maximum execution time for each item is 120s
Hand Grip Dynamometer Strength Tool | 8 months
  It is used in correct position of arm and hand can vary in different grip strength, both for right and left hand will be accessed and scoring start from dominant hand. Interpretation for male in Ib and in( kg), poor in 88-95(Ib) and 40-43kg, average strength 105-114 in (Ib) and 48-51 in( kg) while good strength in 123-141(Ib) and 56-64(kg). and in females values are different poor strength 44-48(ib) and 34-38(kg) , average strength value will be 57-65(ib) and in 26-29 in (kg), while good strength rating is 75-84(ib) and 34-38(kg).
Spinal Cord Independence Measure | 8 months
  There are basically three subscales. First is self care and also for hand function assessment in which 0-4 items and score is 0-20, second is respiration and sphincter management 5-8 items and score is 0-40 while third is mobility with 9-18 items and score is 0-40. Total score is 100 while total items are 19 and assessment completed in 30-45minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, Principal Investigator — Riphah International University
Locations (1):
- Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connor PJ. Prevalence of spinal cord injury in Australia. Spinal Cord. 2005 Jan;43(1):42-6. doi: 10.1038/sj.sc.3101666. PMID 15326472
- [Background] Rahimi-Movaghar V, Saadat S, Rasouli MR, Ganji S, Ghahramani M, Zarei MR, Vaccaro AR. Prevalence of spinal cord injury in Tehran, Iran. J Spinal Cord Med. 2009;32(4):428-31. doi: 10.1080/10790268.2009.11754572. PMID 19777865
- [Background] Jung HY, Lee J, Shin HI. The natural course of passive tenodesis grip in individuals with spinal cord injury with preserved wrist extension power but paralyzed fingers and thumbs. Spinal Cord. 2018 Sep;56(9):900-906. doi: 10.1038/s41393-018-0137-4. Epub 2018 May 22. PMID 29789707
- [Background] Thorsen R, Binda L, Chiaramonte S, Dalla Costa D, Redaelli T, Occhi E, Beghi E, Ferrarin M. Correlation among lesion level, muscle strength and hand function in cervical spinal cord injury. Eur J Phys Rehabil Med. 2014 Feb;50(1):31-8. Epub 2013 Jul 2. PMID 23820875